CLINICAL TRIAL: NCT07358689
Title: Toripalimab Combined With Platinum-based Chemotherapy With or Without H1 Receptor Antagonist (Diphenhydramine) in the Perioperative Treatment of Resectable Non-small Cell Lung Cancer: A Single-center, Randomized Controlled Phase II Clinical Trial
Brief Title: Toripalimab Combined With Platinum-based Chemotherapy With or Without H1 Receptor Antagonist in the Perioperative Treatment of Resectable Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH1RA-NSCLC
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: NSCLC
MeSH Terms: interventions — toripalimab; Diphenhydramine; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tori+D (Experimental): Diphenhydramine combined with Toripalimab plus standard platinum-based chemotherapy as perioperative treatment
  Interventions: Drug: Toripalimab (240mg day1, Q3W*3cycle); Drug: Diphenhydramine; Drug: Platinum-based chemotherapy
- Tori (Other): Toripalimab plus standard platinum-based chemotherapy as perioperative treatment.
  Interventions: Drug: Toripalimab (240mg day1, Q3W*3cycle); Drug: Platinum-based chemotherapy

INTERVENTIONS:
Drug: Toripalimab (240mg day1, Q3W*3cycle) — Toripalimab is a recombinant, humanized programmed death receptor-1 (PD-1) monoclonal antibody that binds to PD-1 and prevents binding of PD-1 with programmed death ligands 1 (PD-L1) and 2 (PD-L2). Toripalimab was administered concurrently with chemotherapy, Q3W
Drug: Diphenhydramine — Diphenhydramine, is an antihistamine. It has antihistamine H1 receptor effects, strong inhibitory effects on the central nervous system, and atropine-like effects. Diphenhydramine was administered 20mg qd IM d0-d2.
  Arms: Tori+D
Drug: Platinum-based chemotherapy — Carboplatin: AUC5 (per Calvert formula); maximum dose: 750 mg；Cisplatin: 75 mg/m² D1, Q3W; Pemetrexed: 500 mg/m² D1, Q3W; Docetaxel: 60-75 mg/m² or Paclitaxel: 175 mg/m², D1, Q3W

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of H1 receptor antagonist (diphenhydramine) combined with toripalimab plus standard platinum-based chemotherapy in the perioperative setting in subjects with operable NSCLC.

The subjects of this study are patients with histologically or cytologically confirmed stage IIIA-IIIB NSCLC (AJCC Version 9) who are planned to receive neoadjuvant therapy with toripalimab combined with standard platinum-based chemotherapy. Eligible subjects were randomized at a 1:1 ratio to receive 3-4 cycles of neoadjuvant diphenhydramine (an H1 receptor antagonist) plus toripalimab and standard platinum-based chemotherapy, or toripalimab plus platinum-based chemotherapy alone, followed by treatment response evaluation and definitive surgery. After surgery, the experimental group will receive maintenance therapy with diphenhydramine (an H1 receptor antagonist) plus toripalimab for 13-14 cycles, while the control group will receive toripalimab monotherapy for the same 13-14 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this study, sign the informed consent form, have good compliance, and are willing to cooperate with follow-up visits;
* Aged 18-75 years, regardless of gender;
* ECOG performance status score of 0-1;
* Expected survival time ≥ 3 months;
* - Pathologically/radiologically confirmed stage IIA-IIIB NSCLC (AJCC 9th Edition). For adenocarcinoma/adenosquamous carcinoma, EGFR wild-type and ALK fusion-negative required before enrollment;
* No prior systemic anti-tumor therapy;
* At least one measurable lesion per RECIST 1.1. Previously irradiated lesions are measurable if progression is confirmed;
* Adequate organ function, as evidenced by meeting the following laboratory parameters:

  1. Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L without administration of granulocyte colony-stimulating factor within the past 14 days;
  2. Platelet count ≥ 80 × 10⁹/L without blood transfusion within the past 14 days;
  3. Hemoglobin > 8 g/dL without blood transfusion or erythropoietin administration within the past 14 days;
  4. Total bilirubin ≤ 1.5 × Upper Limit of Normal (ULN);
  5. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN (for subjects with liver metastasis, AST or ALT ≤ 5 × ULN is acceptable);
  6. Serum creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated by the Cockcroft-Gault formula) ≥ 60 mL/min;
  7. Adequate coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN;
  8. Normal thyroid function, defined as Thyroid Stimulating Hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total triiodothyronine (T3) (or free triiodothyronine [FT3]) and free thyroxine (FT4) within the normal range are also eligible for enrollment;
  9. Myocardial enzyme profile within the normal range;
* Females of childbearing potential: negative pregnancy test (urine/serum) within 3 days pre-first dose (Cycle 1 Day 1); serum test required if urine test unconfirmed. Non-childbearing females: postmenopausal ≥ 1 year, surgically sterile or hysterectomized;
* Subjects at risk of conception: use contraception with annual failure rate < 1% during treatment and 120-180 days post-last dose;

Exclusion Criteria:

* Lung metastases from other primary malignancies;
* Other systemic malignancies (excluding radically treated skin basal/squamous cell carcinoma or resected carcinoma in situ);
* Current or prior myasthenia gravis;
* Current or prior angle-closure glaucoma;
* Current or prior benign prostatic hyperplasia;
* Diphenhydramine allergy;
* Pyloroduodenal obstruction, peptic ulcer-induced pyloric stenosis or bladder neck stenosis;
* Prior radiation therapy meeting any: 1) ≥ 30% bone marrow irradiated within 14 days pre-treatment; 2) Lung lesion radiation > 30 Gy within 6 weeks pre-treatment (must recover from radiation toxicity to Grade ≤ 1, no glucocorticoids, no radiation pneumonitis history);
* Current participation in other interventional clinical studies, or received investigational agents/devices within 4 weeks pre-first dose;
* Systemic anti-lung cancer Chinese patent medicines or immunomodulators (thymosin, interferon, interleukin; excluding local pleural effusion control) within 2 weeks pre-first dose;
* Active autoimmune diseases requiring systemic therapy (disease-modifying drugs, glucocorticoids, immunosuppressants) within 2 years pre-first dose (replacement therapy not considered systemic);
* Ongoing systemic glucocorticoids (excluding topical) or immunosuppressants within 7 days pre-first dose (physiological doses: prednisone ≤ 10 mg/day or equivalent permitted);
* Uncontrolled pleural/peritoneal effusion (eligible if no drainage needed or effusion stable 3 days post-drainage cessation);
* Prior allogeneic organ transplantation (except corneal) or hematopoietic stem cell transplantation;
* Inadequate recovery from prior intervention toxicities/complications (not resolved to Grade ≤ 1 or baseline, excluding fatigue/alopecia);
* Known HIV infection (HIV 1/2 antibody positive);
* Other conditions deemed unsuitable by investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to 1 year

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | Up to 1 year
Overall survival (OS) | Up to 5 years
Objective response rate (ORR) | Up to 1 year
Event-free survival (EFS) | Up to 5 years
Incidence of Treatment-Related Adverse Events | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China